CLINICAL TRIAL: NCT04382989
Title: The Influence of Various Maternal, Infant and Environmental Factors on Human Milk Composition Among Lithuanian Women
Brief Title: Factors Influencing the Composition of Human Milk
Status: Completed | Type: Observational
Sponsor: Vilnius University (Other)
Collaborators: University of Cagliari (Other)
Responsible Party: Sponsor
Other Study IDs: MPS-2017
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Breast Milk Collection
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Mothers of extremely preterm infants: (gestational age < 28 weeks)
  Interventions: Device: Analysis of human milk composition by mid-infrared spectrophotometry
- Mothers of very preterm infants: (gestational age 28 - 31 weeks)
  Interventions: Device: Analysis of human milk composition by mid-infrared spectrophotometry
- Mothers of moderate and late preterm infants: (gestational age 32 - 36 weeks)
  Interventions: Device: Analysis of human milk composition by mid-infrared spectrophotometry
- Mothers of term infants: (gestational age ≥ 37 weeks)
  Interventions: Device: Analysis of human milk composition by mid-infrared spectrophotometry

INTERVENTIONS:
Device: Analysis of human milk composition by mid-infrared spectrophotometry — Analysis of human milk macronutrient content was performed by mid-infrared spectrophotometry using a Miris Human Milk Analyser.
  An immune-enzymatic ELISA assays were used to estimate lysozyme and lactoferrin concentrations in human milk.
  Other Names: Holder pasteurisation

SUMMARY:
This study aims for characterization of different maternal, infant and environmental factors (e.g. maternal age, pregnancy duration, lactation period, baby gender, circadian rhythm, Holder pasteurisation, etc.) that influence human milk composition.

DETAILED DESCRIPTION:
The study consists of three parts. In the first part the investigators aim to evaluate human milk macronutrient composition depending on the time after delivery and pregnancy duration.

In the second part the investigators aim to evaluate the circadian variation of human milk macronutrient and energy content depending on pregnancy duration.

In the third part the investigators aim to evaluate the influence of Holder pasteurisation on human milk macronutrient, metabolome and bioactive protein (lysozyme and lactoferrin) content.

ELIGIBILITY:
Inclusion Criteria:

having obtained informed consent; after a single-birth pregnancy; women who were not on a special diet; lactating mothers who could not breastfeed their newborns due to the baby's medical condition (either prematurity or disease) but who expressed milk.

-

Exclusion Criteria:

breastfeeding mothers; history of maternal diabetes, hepatitis B or C, HIV, tuberculosis, mastitis, or oncological disease; drug addicted.

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Lactating women
Study Population: Mothers of newborns admitted at Neonatal Center of Vilnius University Hospital Santaros Klinikos, Lithuania
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Quantification of total protein concentration in human milk | from the 2nd week, up to 2 months after delivery
  Mid-infrared spectrophotometry

SECONDARY OUTCOMES:
Quantification of total lipids and carbohydrate in human milk | from the 2nd week, up to 2 months after delivery
  Mid-infrared spectrophotometry
Quantification of lactoferrin in human milk | 14-16 days after delivery
  An immune-enzymatic ELISA assay
Quantification of lysozyme in human milk | 14-16 days after delivery
  An immune-enzymatic ELISA assay
Human milk metabolome analysis | 15-17 days after delivery
  Nuclear Magnetic Resonance (NMR) analysis

CONTACTS AND LOCATIONS:
Overall Officials: Vytautas Usonis, MD, Study Director — Vilnius University
Locations (1):
- Neonatal centre of Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paulaviciene IJ, Liubsys A, Eidukaite A, Molyte A, Tamuliene L, Usonis V. The Effect of Prolonged Freezing and Holder Pasteurization on the Macronutrient and Bioactive Protein Compositions of Human Milk. Breastfeed Med. 2020 Sep;15(9):583-588. doi: 10.1089/bfm.2020.0219. Epub 2020 Aug 26. PMID 32856945